CLINICAL TRIAL: NCT01043705
Title: Centurion and Citadel Studies of TYRX™ Anti-Bacterial Envelope and Custom Mesh for Prevention of Infection Following CIED Replacement With a CRT or ICD
Brief Title: TYRX™ Envelope for Prevention of Infection Following Replacement With a CRT or ICD
Acronym: Centurion
Status: Completed | Type: Observational
Sponsor: TYRX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-2009-2; NCT01043861 (obsolete NCT alias)
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Results first posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-10

CONDITIONS: Cardiac Implantable Electronic Device Infection
Keywords: Pacemaker infection; Defibrillator infection; ICD infection; CRT infection; Cardiovascular implantable electronic device infection; Infection; Pacemaker, Artificial; Defibrillators
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- CIED replacement with CRT and TYRX: (Prospective Arm) Patients who have undergone CIED replacement with a CRT and the TYRX Anti-bacterial envelope, with or without lead revision.
- CIED replacement with ICD and TYRX: (Prospective Arm) Patients who have undergone CIED replacement with an ICD and the TYRX Anti-bacterial envelope, with or without lead revision.
- CIED replacement with ICD or CRT and TYRX: (Prospective Arm) Patients who have undergone CIED replacement with an ICD or CRT and the TYRX Anti-bacterial envelope, with or without lead revision.
- CIED replacement w/ CRT & no TYRX: (Retrospective Case-Control Arm) Patients who have undergone CIED replacement with a CRT and no TYRX Anti-bacterial envelope, with or without lead revision/addition.
- CIED replacement w/ CRT & TYRX vs. Case Match Arm: Patients who have undergone CIED replacement with a CRT and TYRX Anti-bacterial envelope, with or without lead revision/addition. Cohort is TYRX Case, Matched to Retrospective Case-Control Arm)

SUMMARY:
The purpose of this study is to compare the incidence of cardiac implantable electronic device (CIED) infection and CIED mechanical complication after CIED replacement with a high-power cardiac implantable electronic device; either a cardiac resynchronization therapy device (CRT), or an implantable cardioverter defibrilator (ICD) and TYRX Anti-Bacterial Envelope (formerly known as "AIGISRx"), to the incidence, after replacement with an ICD or CRT and no TYRX.

DETAILED DESCRIPTION:
Cardiac implantable electronic device (CIED) infection is associated with significant morbidity and expense. The frequency of CIED infection is increasing faster than the frequency of CIED implants, suggesting more effective prophylactic strategies are needed.

The TYRX Anti-Bacterial Envelope is an FDA-cleared polypropylene mesh that is intended to securely hold a pacemaker pulse generator or defibrillator (ICD) in order to create a stable environment when implanted in the body. It contains the antimicrobial agents, rifampin and minocycline, which have been shown to reduce infection in an in vivo model of bacterial contamination following surgical implant of the generator or defibrillator.

This is a prospective, observational, multicenter registry of subjects undergoing CIED replacement with an ICD or CRT and TYRX, with or without lead revision/addition. The registry subjects will be compared to a published historical control group undergoing CIED replacement with an ICD or CRT and no TYRX , with or without lead revision/addition. The CRT registry subjects will also be compared to a case-matched retrospective control group undergoing CIED replacement with a CRT and no TYRX , with or without lead revision/addition. The primary study endpoints are major CIED infection and CIED mechanical complication during the 12 months following CIED replacement with an ICD or CRT.

Originally executed as two separate studies (Citadel - ICDs) and (Centurion - CRTs), a protocol amendment was executed in 2012 due to slow enrollment, combining the databases for analysis of results.

ELIGIBILITY:
Inclusion Criteria: - Prospective Arms

* Qualifying CIED Implant procedure was replacement with an ICD or CRT and TYRX, with or without lead revision/addition
* Received a complete TYRX Anti-Bacterial Envelope Model# 3122 or #3133 according to the Instructions for Use (IFU)
* Clinically stable to tolerate procedure
* 18 years or older
* Able to return for follow-up care through the 12-month visit, or able to have referring physician provide follow-up data to study site by telephone

Exclusion Criteria: - Prospective Arm

* Unable/unwilling to provide informed consent
* Contraindication to receiving the TYRX device, in accordance with the package labeling
* Pregnant or was at risk for becoming pregnant in the 30 day period following the Qualifying TYRX Implant
* Current CIED infection, or the indication for Qualifying CIED Implant was replacement of CIED that was explanted for infection
* Clinical diagnosis of an active infection at the time of CIED implant, including pneumonia, urinary tract infection, endovascular, cellulitis, bacteremia, or other major systemic infection. (Note: asymptomatic bacteremia without UTI is not an exclusion criterion)
* Generator replacement required planned lead extraction
* Participating in another clinical study evaluating a drug or device designed to reduce CIED infections
* Life expectancy of less than 6 months
* Expected to receive a heart transplant within 6 months
* With the exception of the elderly in good mental health, all vulnerable subjects as defined by the FDA Office of Human Research Protection or local IRB will be excluded

Inclusion Criteria: - Case-matched retrospective Control Arm

* Qualifying CIED Implant was replacement with a CRT and TYRX, with or without lead revision/addition
* First un-enrolled patient meeting case-matching criteria in series of patients implanted with a CIED and no TYRX beginning 24 months prior to the date of first TYRX implant at site. If no matching patients in this period, first un-enrolled matching patient implanted with a CIED and no TYRX beginning 24 months prior to the first TYRX implant at site, searching in reverse chronological order
* Had at least one of following by date of enrollment into the study:

  1. ≥ 12 months follow-up after Qualifying TYRX Implant
  2. Subsequent TYRX Procedure that required opening the generator pocket or implant incision ≤ 12 months after Qualifying TYRX Implant (e.g. battery change, upgrade, lead revision, explant)
  3. Death ≤ 12 months after Qualifying CIED Implant
* Survived Qualifying CIED Implant to discharge, died of a CIED infection or Mechanical Complication prior to hospital discharge, or died for any reason un-related to Qualifying CIED Implant prior to hospital discharge
* 18 years or older

Exclusion Criteria: - Case-matched retrospective Control Arm

* Contraindication to receiving the TYRX device, in accordance with the package labeling
* Pregnant or became pregnant in the 30 day period following the Qualifying TYRX Implant.
* CIED infection, or the indication for Qualifying CIED Implant was replacement of CIED that was explanted for infection
* Clinical diagnosis of an active infection at the time of Qualifying CIED Implant, including pneumonia, urinary tract infection, endovascular, cellulitis, bacteremia, or other major systemic infection (Note: asymptomatic bacteriuria without UTI is not an exclusion criterion)
* Lead extraction was performed at the Qualifying CIED Implant
* Participated in another clinical study evaluating a drug or device intended to reduce CIED infections
* Received a heart transplant within 6 months of Qualifying CIED Implant
* With the exception of the elderly in good mental health, all vulnerable subjects as defined by the FDA Office of Human Research Protection or local IRB will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone CIED replacement with an ICD or CRT, with or without (CRT retrospective group only) an TYRX Anti-bacterial Envelope, at US medical centers.
Sampling Method: Non-Probability Sample
Enrollment: 1262 (Actual)
Dates: Start 2010-01; Primary Completion 2014-07 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (52):
- United States (52):
  - Princeton Medical Center, Birmingham, Alabama
  - Decatur General Hospital, Decatur, Alabama
  - Eliza Coffee Memorial Hospital, Florence, Alabama
  - Riverview Regional Hospital, Gadsden, Alabama
  - Arizona Heart Hospital, Scottsdate, Arizona
  - Community Memorial Hospital, Ventura, California
  - Watsonville Community Hospital, Watsonville, California
  - Citrus Memorial Hospital, Inverness, Florida
  - Osceola Regional Medical Center, Kissimmee, Florida
  - University of Miami, Miami, Florida
  - Orlando Regional Hospital, Orlando, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Piedmont Medical Center, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Veteran's Administration Medical Center, Atlanta, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Trinity Medical Center, Rock Island, Illinois
  - St. John's Hospital, Springfield, Illinois
  - St. Mary's Medical, Hobart, Indiana
  - Community Hospital, Munster, Munster, Indiana
  - St. Margaret Mercy, Munster, Indiana
  - P and S Surgical Hospital, Monroe, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Penninsula Regional Medical Center, Salisbury, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Gulfport Memorial Hospital, Biloxi, Mississippi
  - Keesler Air Force Base Hospital, Biloxi, Mississippi
  - Southern Heart Center, Hattiesburg, Mississippi
  - Alegent Health, Omaha, Nebraska
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - St. Francis Hospital, Hamilton, New Jersey
  - Newark Beth Israel Hospital, Newark, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Our Lady of Lourdes Hospital, Sewell, New Jersey
  - St. Luke's - Roosevelt Hospital, New York, New York
  - Frye Regional Medical Center, Hickory, North Carolina
  - Catholic Health Partners, Youngstown, Ohio
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Pinnacle Health Harrisburg Hospital, Harrisburg, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Landmark Medical Center, Woonsocket, Rhode Island
  - Stern Cardiovascular Foundation, Germantown, Tennessee
  - University of Tenn. Medical Center - Knoxville, Knoxville, Tennessee
  - Texas Heart Institute - St. Luke's Episcopal Hospital, Houston, Texas
  - NE Methodist, San Antonio, Texas
  - Aurora Health Care, Milwaukee, Wisconsin

REFERENCES:
- [Background] Sohail MR, Henrikson CA, Braid-Forbes MJ, Forbes KF, Lerner DJ. Comparison of mortality in women versus men with infections involving cardiovascular implantable electronic device. Am J Cardiol. 2013 Nov 1;112(9):1403-9. doi: 10.1016/j.amjcard.2013.06.031. Epub 2013 Aug 22. PMID 23972346
- [Background] Ballo P, Chiodi L, Zuppiroli A. Cardiac implantable electronic devices: prevention starts from ethics. Arch Intern Med. 2012 Apr 23;172(8):670-1; author reply 671-2. doi: 10.1001/archinternmed.2012.346. No abstract available. PMID 22529239
- [Derived] Henrikson CA, Sohail MR, Acosta H, Johnson EE, Rosenthal L, Pachulski R, Dan D, Paladino W, Khairallah FS, Gleed K, Hanna I, Cheng A, Lexcen DR, Simons GR. Antibacterial Envelope Is Associated With Low Infection Rates After Implantable Cardioverter-Defibrillator and Cardiac Resynchronization Therapy Device Replacement: Results of the Citadel and Centurion Studies. JACC Clin Electrophysiol. 2017 Oct;3(10):1158-1167. doi: 10.1016/j.jacep.2017.02.016. Epub 2017 May 31. PMID 29759500

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Enrolled = 1 January 2010; Last Patient Enrolled = 7 May 2013
Pre-assignment Details: CRT and ICD Implant patients with TYRX Implant; Full analysis cohort = 1,129 patients. 670 patient CRT + TYRX cohort is subset. 459 patient ICD + TYRX is subset. 578 CRT+ TYRX patient cohort is subset matched to 578 patient CRT/no TYRX retrospective patient arm.
Groups:
- ICD With TYRX Implant: All patients receiving a TYRX envelope who were eligible to participate having a replacement ICD implant
- CRT and TYRX Cases, Matched to Retrospective Non-TYRX Implants: Patients receiving a TYRX envelope who were eligible to participate having a replacement CRT implant who have a valid non-TYRX implant case-match
- CRT With no TYRX Retrospective Case Control: Retrospective site matched and case-matched CRT replacement patients who did not receive a TYRX envelope selected in the era just prior to availability of TYRX Envelope
Period: Overall Study
Arm/Group | ICD With TYRX Implant | CRT and TYRX Cases, Matched to Retrospective Non-TYRX Implants | CRT With no TYRX Retrospective Case Control
Started | 459 | 578 | 578
Completed | 352 | 447 | 498
Not Completed | 107 | 131 | 80
Not completed — Death | 28 | 60 | 26
Not completed — Lost to Follow-up | 27 | 12 | 0
Not completed — Multiple Reasons | 4 | 7 | 0
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Withdrawal by Subject | 8 | 6 | 0
Not completed — Site Closure | 8 | 0 | 0
Not completed — Subsequent Procedure | 9 | 24 | 29
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Screen Fail | 21 | 0 | 0
Not completed — Other | 0 | 19 | 25

BASELINE CHARACTERISTICS:
Population: Prospective Population: ICD and CRT replacement implant patients receiving a TYRX Envelope Retrospective Population: CRT Patients receiving a CRT and no TYRX envelope. Patients are site medical charts from just previous to use of TYRX Evelope
Groups:
- CIED Replacement With CRT and no TYRX: (Retrospective Case-Control Arm) Patients who have undergone CIED replacement with a CRT and no TYRX Anti-bacterial envelope, with or without lead revision/addition.
- CIED Replacement With CRT and TYRX Vs. Case Match Arm: Prospective CRT patients who received a TYRX envelope and had a valid case match retrospective patient. This is a subset of all CRT/TYRX patients
- Total: Total of all reporting groups
Arm/Group | CIED Replacement With ICD and TYRX | CIED Replacement With CRT and no TYRX | CIED Replacement With CRT and TYRX Vs. Case Match Arm | Total
Number analyzed (Participants) | 459 | 578 | 578 | 1615
Age, Continuous [Median (Standard Deviation); unit: Years] | 70 (12.01) | 73 (10.94) | 73 (10.70) | 72 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 339 | 434 | 444 | 1217
  Male | 120 | 144 | 134 | 398

OUTCOME MEASURES:

1. Primary Outcome: Major CIED Infection
Description: CIED Major Infections
Time Frame: 12 months
Population: Evaluable patients that have valid entry criteria
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Groups:
- CIED Replacement With CRT and TYRX vs. Case Match Arm: CIED replacement with CRT and TYRX vs. Case Match Arm; CRT patients who have corresponding non-TYRX implant case-match
Arm/Group | CIED Replacement With CRT and TYRX | CIED Replacement With CRT and no TYRX | CIED Replacement With CRT and TYRX vs. Case Match Arm
Number analyzed (Participants) | 670 | 578 | 578
percentage of Participants | 0.6 [0 to 1.4] | 1.0 [0 to 2.0] | 0.7 [0 to 1.6]
Statistical Analysis 1: Comparison: CIED Replacement With CRT and TYRX vs CIED Replacement With CRT and no TYRX; Test type: Superiority or Other; p = 0.0023, Fisher Exact; One sided Fisher's exact test. = 0.0044, 95% CI 1-sided [upper limit 0.009]
Statistical Analysis 2: Comparison: CIED Replacement With CRT and TYRX vs CIED Replacement With CRT and no TYRX; Test type: Superiority or Other; p = 0.0052, Fisher Exact; 1-sided Fisher's Exact Text = 0.002, 95% CI 1-sided [upper limit 0.01]
Statistical Analysis 3: Comparison: CIED Replacement With CRT and TYRX; Test type: Superiority or Other; p = 0.0176, Fisher Exact; 1-sided Fisher's Exact Test = 0.006, 95% CI 1-sided [upper limit 0.014]
Statistical Analysis 4: Comparison: CIED Replacement With CRT and no TYRX vs CIED Replacement With CRT and TYRX vs. Case Match Arm; Test type: Superiority or Other; p = 0.3764, Fisher Exact; Fisher's Exact Test = .7

2. Primary Outcome: CIED Mechanical Complication
Description: All mechanical Complications related to CIED Implant
Time Frame: 12 months
Population: TYRX implants vs. published comparator are "prospective arm" patients. Non-TYRX CIED retrospective arm vs. TYRX CIED replacements are nested, case-control cohort.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | CIED Replacement With ICD and TYRX | CIED Replacement With CRT and no TYRX | CIED Replacement With CRT and TYRX vs. Case Match Arm
Number analyzed (Participants) | 459 | 578 | 578
percentage of Participants | 3.1 [1.7 to 5.1] | 5.5 [3.8 to 7.7] | 5.4 [3.7 to 7.5]
Statistical Analysis 1: Comparison: CIED Replacement With ICD and TYRX vs CIED Replacement With CRT and no TYRX; Test type: Superiority or Other; p = 0.0005, 1-sided Chi-square; Rate compared to performance goal = 4.4, 95% CI 2-sided [3.3 to 5.8]
Statistical Analysis 2: Comparison: CIED Replacement With ICD and TYRX; Test type: Superiority or Other; p = 0.0444, 1-sided Chi-square test; Rate compared to a performance goal = 3.1, 95% CI 2-sided [1.7 to 5.1]
Statistical Analysis 3: Comparison: CIED Replacement With ICD and TYRX vs CIED Replacement With CRT and no TYRX; All types of mechanical complications combined; Test type: Superiority or Other; p = 0.0006, 1-sided Chi-squared test; rate compared to performance goal = 5.4, 95% CI 2-sided [3.8 to 5.4]
Statistical Analysis 4: Comparison: CIED Replacement With CRT and no TYRX vs CIED Replacement With CRT and TYRX vs. Case Match Arm; All mechanical complications, retrospective, non-TYRX cohort; Test type: Superiority or Other; p = 0.0745, Chi-squared; Descriptive = 5.4, 95% CI 2-sided [3.7 to 7.5]

ADVERSE EVENTS:
Time Frame: During 12 month follow up period
Description: Note that non-serious adverse events were not collected or assessed as part of this study.
  Adverse events coded as "death" do not have further description.
Arm/Group | CIED Replacement With CRT and TYRX | CIED Replacement With ICD and TYRX
Serious Adverse Events (participants affected / at risk) | 96/578 | 46/459
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CIED Replacement With CRT and TYRX (N=578) | CIED Replacement With ICD and TYRX (N=459)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 2 (2) | 1 (1)
Aortic Valve Stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Atrial Thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Amyloidosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 5 (5) | 2 (2)
Cardiac disorder (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac Failure Acute (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 18 (18) | 6 (6)
Cardio-respiratory failure (Cardiac disorders) | 4 (4) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 1 (1)
Cardiopulmonary Failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 3 (3) | 0 (0)
Ischemic Cardiomyopathy (Cardiac disorders) | 3 (3) | 0 (0)
Low Cardiac Output Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Mitral Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Restrictive Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Tricuspid Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Gastrointestinal Heamorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse Drug Reaction (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0)
Brain Death (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Complication of Device Removal (General disorders) | 0 (0) | 1 (1)
Condition Aggravated (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 45 (45) | 24 (24)
Device Component Issue (General disorders) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 4 (4) | 1 (1)
Device Electrical Finding (General disorders) | 0 (0) | 1 (1)
Device Failure (General disorders) | 0 (0) | 1 (1)
Device Lead Damage (General disorders) | 2 (2) | 1 (1)
Device Lead Issue (General disorders) | 0 (0) | 1 (1)
Device Malfunction (General disorders) | 1 (1) | 1 (1)
Device Pacing Issue (General disorders) | 0 (0) | 1 (1)
Device Stimulation Issue (General disorders) | 1 (1) | 0 (0)
Feeling Hot (General disorders) | 1 (1) | 0 (0)
General Physical Health Deterioration (General disorders) | 4 (4) | 1 (1)
Impaired Healing (General disorders) | 1 (1) | 0 (0)
Implant Site Discharge (General disorders) | 1 (1) | 0 (0)
Implant Site Haematoma (General disorders) | 6 (6) | 0 (0)
Implant Site Haemorrhage (General disorders) | 0 (0) | 1 (1)
Implant Site Pain (General disorders) | 0 (0) | 1 (1)
Medical Device Site Reaction (General disorders) | 1 (1) | 0 (0)
Multi-Organ Failure (General disorders) | 1 (1) | 0 (0)
Multimorbidity (General disorders) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Treatment Failure (General disorders) | 1 (1) | 0 (0)
Cardiac Valve Vegetation (Infections and infestations) | 1 (1) | 0 (0)
Device Related Infection (Infections and infestations) | 2 (2) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Implant Site Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Implant Site Infection (Infections and infestations) | 2 (2) | 3 (3)
Infected Skin Ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (7) | 2 (2)
Pneumonia Staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Septic Shock (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Eschar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision Site Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Blood Creatinine Increased (Investigations) | 1 (1) | 1 (1)
Blood Culture Positive (Investigations) | 1 (1) | 0 (0)
Blood Urea Increased (Investigations) | 1 (1) | 0 (0)
Blood Urea Nitrogen/Creatinine Ratio Increased (Investigations) | 1 (1) | 0 (0)
International Normalised Ratio Increased (Investigations) | 1 (1) | 0 (0)
Troponin Increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to Thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Hodgin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Small Cell Lung Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 2 (2) | 0 (0)
Loss of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 2 (2) | 0 (0)
Renal Failure (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal Failure Acute (Renal and urinary disorders) | 4 (4) | 0 (0)
Renal Failure Chronic (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal Mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung Consolidation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Long Disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic Valve Replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac Pacemaker Removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac Pacemaker Replacement (Surgical and medical procedures) | 3 (3) | 1 (1)
Cardio Pacemaker Revision (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardioversion (Surgical and medical procedures) | 2 (2) | 1 (1)
Chest Tube Insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Drain Placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Emergency Care (Surgical and medical procedures) | 5 (5) | 1 (1)
Endotracheal Intubation (Surgical and medical procedures) | 1 (1) | 0 (0)
Haemodialysis (Surgical and medical procedures) | 1 (1) | 1 (1)
Hospice Care (Surgical and medical procedures) | 4 (4) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 27 (27) | 10 (10)
Implantable Defibrillator Insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Incisional Drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Mechanical Ventilation (Surgical and medical procedures) | 1 (1) | 0 (0)
Medical Device Change (Surgical and medical procedures) | 1 (1) | 0 (0)
Medical Device Removal (Surgical and medical procedures) | 1 (1) | 1 (1)
Packed Red Blood Cell Transfusion (Surgical and medical procedures) | 1 (1) | 0 (0)
Palliative Care (Surgical and medical procedures) | 2 (2) | 3 (3)
Rehabilitation Therapy (Surgical and medical procedures) | 1 (1) | 1 (1)
Tracheostomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Ventricular Assist Device Insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Withdrawal of Life Support (Surgical and medical procedures) | 1 (1) | 0 (0)
Wound Drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Distributive Shock (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This was a non-randomized study and did not have an active comparator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No